CLINICAL TRIAL: NCT07070219
Title: A Single-Arm, Open-Label, Multi-Center, Phase 1b/ 2 Study to Evaluate the Safety, Efficacy, and Cellular Pharmacokinetic Profile of CTD402 in Participants With Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL) and Lymphoblastic Lymphoma (T-LBL) (TENACITY-01)
Brief Title: A Study of CTD402 in T-ALL/LBL Patients
Acronym: TENACITY-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BIOHENG THERAPEUTICS US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-CTD402-201
Record Dates: First submitted 2025-07-07; First posted 2025-07-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphocytic Leukemia Refractory; Lymphoma, Lymphoblastic
Keywords: CAR-T Therapy; relapsed/refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CTD402 Cell Infusion (Experimental)
  Interventions: Drug: CTD402 CAR T Cell Injection

INTERVENTIONS:
Drug: CTD402 CAR T Cell Injection — CAR T cells

SUMMARY:
The goal of the TENACITY-01 clinical trial is to learn if CTD402 UCART is safe and effective for relapsed/refractory T-ALL/LBL patients.

Participants with relapsed/refractory T-ALL/LBL over the age of 12 will be eligible to participate.

Participants will receive one infusion of CTD402 on Day 0 and will be evaluated for anti-tumor activity by an independent review committee based on the NCCN criteria for T-ALL and the Lugano 2014 criteria for T-LBL.

Patients will be followed for up to 24 months in this study and will be required to enroll under a separate long term follow up protocol to be followed for up to 15 years.

DETAILED DESCRIPTION:
TENACITY-01 is a single-arm, open-label, multi-center, Phase 1b/2 study to assess the safety and efficacy of CTD402 in adolescent (≥ 12 to 17 years) and adult participants with relapsed/refractory (r/r) T-ALL/LBL. Approximately 18 participants will be enrolled in the Phase 1b portion of the study to evaluate the safety and establish the RP2D of CTD402, with approximately 18 participants receiving CTD402 at RP2D. Approximately 36 participants will be enrolled in the Phase 2 portion of the study to further confirm the efficacy and safety of CTD402.

Both the phase 1b and phase 2 portions will consist of the following sequential phases: screening (up to 2 weeks), lymphodepletion period (within 7 days prior to treatment), CTD402 treatment (a single dose), primary follow-up period (up to 2 years). Once a participant receives the first dose of lymphodepleting chemotherapy regimen, the participant will be considered enrolled into the study.

Long term follow-up will be conducted under a separate protocol until 15 years following CTD402 infusion for survival, toxicity, RCR monitoring, and secondary malignancy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, ≥ 12 years of age.
2. Participants with body weight ≥ 40 kilogram.
3. Relapsed or refractory T-ALL/LBL is defined as one of the following:

   1. Relapsed or refractory disease after two or more lines of systemic therapy;
   2. The first relapse occurs within 12 months after first remission;
   3. Relapse after allogeneic HSCT and must be ≥100 days from HSCT prior to screening period.
4. The presence of bone marrow lymphoblasts is ≥ 5% as determined by morphologic evaluation or evidence of extramedullary disease at screening.
5. Have eligible HLA-matched related donor (MRD) or unrelated donor (URD), eligible haploidentical donor (HID) or syngeneic donors.
6. Adequate organ function
7. Karnofsky PS ≥ 60 (for participants age ≥ 16) or Lansky PS ≥ 60 (for participants < 16) at screening.

Key Exclusion Criteria:

1. Participants with concomitant genetic syndromes associated with bone marrow failure states or any other known bone marrow failure syndrome.
2. Active central nervous system (CNS) involvement
3. Participants with following cardiac conditions will be excluded:

   1. History of heart failure New York Heart Association (NYHA) class III or IV;
   2. History of myocardial infarction, cardiovascular angioplasty or stenting, unstable angina, or other serious heart diseases within 12 months of enrollment.
4. Primary immune deficiency.
5. Presence of uncontrolled infections.
6. Known history of infection with the human immunodeficiency virus (HIV); hepatitis C virus and syphilis.
7. Active or latent hepatitis B virus infection
8. Epstein-Barr virus (EBV), Cytomegalovirus (CMV) DNA or IgM positive at screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety Profile | 24 months
  Incidence of dose limiting toxicities including incidence of adverse events and graft vs host disease
Response Evaluation | 24 months
  Percentage of participants who achieve overall complete remission (OCR) assess by an independent review committee

SECONDARY OUTCOMES:
Characterize the cPK profile of CTD402 | 24 months
  CTD402 cellular pharmacokinetic (PK)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - Sarah Cannon Research Insitute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No